CLINICAL TRIAL: NCT04882540
Title: An Open-label, Single-arm Study to Evaluate the Pharmacokinetics and Safety of a Single and Multiple Oral Doses of Brivaracetam in Healthy Adult Chinese Subjects
Brief Title: A Study to Evaluate the Pharmacokinetics and Safety of Brivaracetam in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EP0101
Record Dates: First submitted 2021-05-06; First posted 2021-05-12 (Actual); Results first posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2022-05

CONDITIONS: Healthy Participants
Keywords: Epilepsy; Healthy participants; Phase 1; Brivaracetam
MeSH Terms: conditions — Epilepsy | interventions — brivaracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- brivaracetam (Experimental): This is a Single-Arm study with Single- and Multiple- Dose Periods. Study participants will receive a single dose of brivaracetam (BRV) on Day 1 and will then receive multiple doses of brivaracetam from Day 5-10.
  Interventions: Drug: brivaracetam

INTERVENTIONS:
Drug: brivaracetam — * Pharmaceutical form: Film-coated tablets
  * Concentration: 100 mg tablets
  * Route of administration: Oral use
  Other Names: Briviact

SUMMARY:
The purpose of the study is to assess the pharmacokinetics, safety, and tolerability of brivaracetam after a single dose and multiple doses in healthy adult Chinese Study Participants.

ELIGIBILITY:
Inclusion Criteria:

* An Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved written Informed Consent form is signed and dated by the subject
* Subject is considered reliable and capable of adhering to the protocol (eg, able to understand and complete diaries), visit schedule, or medication intake according to the judgment of the Investigator
* Subjects are Chinese males and females born in China between 18 and 45 years of age (both inclusive) whose parents are of Chinese origin
* Subjects with body mass index (BMI) from 19 to 24 kg/m^2 (both inclusive). Minimum body weight is equal to or more than 50 kg
* Subjects with supine blood pressure levels of between 90 to 150 and 60 to 90 mmHg (inclusive) for systolic and diastolic, respectively, with pulse rate of 50 to 100 beats per minute (bpm) (supine position, inclusive) at Screening Visit
* Subjects without clinically relevant abnormalities in a standard 12-lead Electrocardiogram (ECG) at Screening Visit judged by the Investigators
* Subjects with laboratory values within the reference range at Screening Visit, or those with values exceeding the reference range but judged by the Investigators to be not clinically significant to their participation in the study

Exclusion Criteria:

* Subject has participated in another study of an investigational medicinal product (IMP) (or a medical device) within the previous 30 days or is currently participating in another study of an IMP (or a medical device)
* Subject has any medical or psychiatric condition that, in the opinion of the Investigator, could jeopardize or would compromise the subject's ability to participate in this study
* Pregnant, lactating, or sexually active women with childbearing potential who are not using a medically accepted birth control method
* Subject has a known hypersensitivity to any components of the IMP or any of its excipients
* Subjects with any previous or current cardiovascular, respiratory, hepatic, renal, digestive, endocrine, or nervous system disorder that may affect absorption, secretion, metabolism, or excretion of the investigational product per Investigator judgement
* Subjects showing a positive result for hepatitis B surface antigen, hepatitis C virus antibody, human immunodeficiency virus antibody, or syphilis test at Screening Visit

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2021-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (1):
- Ep0101 101, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, IPD cannot be adequately anonymized i.e., there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial cannot be shared.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll study participants in May 2021 and concluded in June 2021.
Pre-assignment Details: Participant Flow refers to the Safety Set.
Groups:
- Brivaracetam: Participants received a single dose of brivaracetam (BRV) 100 milligrams (mg), orally on Day 1 in the single dose period and received BRV 200 mg/day, orally from Day 5 to 9 and 100 mg on Day 10 in the multiple dose period.
Period: Overall Study
Arm/Group | Brivaracetam
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The Safety Set consisted of all participants who received at least 1 dose of BRV.
Groups:
- Brivaracetam: Participants received a single dose of BRV 100 mg, orally on Day 1 in the single dose period and received BRV 200 mg/day, orally from Day 5 to 9 and 100 mg on Day 10 in the multiple dose period.
Arm/Group | Brivaracetam
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.9 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 12

OUTCOME MEASURES:

1. Primary Outcome: Plasma Concentration of BRV and Its Metabolites (Ucb-42145, Ucb-100406-1, ucb107092-1) After Single Dose
Time Frame: Day 1: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, and 72 hours postdose
Population: The PK-PPS consisted of all participants who were included in the safety set and also had a sufficient number of bioanalytical assessments to calculate reliable estimates for the primary PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Groups:
- Brivaracetam: Participants received a single dose of BRV 100 mg, orally on Day 1 in the single dose period.
Arm/Group | Brivaracetam
Number analyzed (Participants) | 12
nanograms/milliliter (ng/mL)
  BRV- Day 1: Predose | NA (NA) — Means, standard deviation (SDs) and coefficient of variation (CVs) were only calculated if at least 2/3 of the concentrations are above lower limit of quantification (LLOQ).
  BRV- Day 1: 0.25 hour postdose | 1039 (134)
  BRV- Day 1: 0.50 hour postdose | 2610 (46.2)
  BRV- Day 1: 1 hour postdose | 2725 (19.6)
  BRV- Day 1: 1.5 hours postdose | 2458 (15.9)
  BRV- Day 1: 2 hours postdose | 2602 (18.2)
  BRV- Day 1: 3 hours postdose | 2387 (21.3)
  BRV- Day 1: 4 hours postdose | 2181 (22.8)
  BRV- Day 1: 6 hours postdose | 1793 (22.4)
  BRV- Day 1: 9 hours postdose | 1389 (27.8)
  BRV- Day 1: 12 hours postdose | 1064 (28.8)
  BRV- Day 1: 16 hours postdose | 747.7 (32.7)
  BRV- Day 1: 24 hours postdose | 423.8 (45.9)
  BRV- Day 1: 36 hours postdose | 157.6 (64.4)
  BRV- Day 1: 48 hours postdose | 68.75 (86.6)
  BRV- Day 1: 72 hours postdose | 9.372 (229)
  ucb-42145- Day 1: Predose | NA (NA) — Means, SDs and CVs were only calculated if at least 2/3 of the concentrations are above LLOQ.
  ucb-42145- Day 1: 0.25 hour postdose | 4.480 (131)
  ucb-42145- Day 1: 0.50 hour postdose | 27.48 (66.8)
  ucb-42145- Day 1: 1 hour postdose | 78.18 (31.8)
  ucb-42145- Day 1: 1.5 hours postdose | 130.5 (19.6)
  ucb-42145- Day 1: 2 hours postdose | 155.9 (22.8)
  ucb-42145- Day 1: 3 hours postdose | 187.8 (30.3)
  ucb-42145- Day 1: 4 hours postdose | 149.4 (21.8)
  ucb-42145- Day 1: 6 hours postdose | 122.5 (16.5)
  ucb-42145- Day 1: 9 hours postdose | 112.6 (25.0)
  ucb-42145- Day 1: 12 hours postdose | 75.73 (26.3)
  ucb-42145- Day 1: 16 hours postdose | 59.17 (26.6)
  ucb-42145- Day 1: 24 hours postdose | 37.46 (38.4)
  ucb-42145- Day 1: 36 hours postdose | 12.82 (50.8)
  ucb-42145- Day 1: 48 hours postdose | 6.222 (64.1)
  ucb-42145- Day 1: 72 hours postdose | NA (NA) — Means, SDs and CVs were only calculated if at least 2/3 of the concentrations are above LLOQ.
  ucb-100406-1- Day 1: Predose | NA (NA) — Means, SDs and CVs were only calculated if at least 2/3 of the concentrations are above LLOQ.
  ucb-100406-1- Day 1: 0.25 hour postdose | 7.364 (146)
  ucb-100406-1- Day 1: 0.5 hour postdose | 29.78 (88.5)
  ucb-100406-1- Day 1: 1 hour postdose | 39.97 (81.2)
  ucb-100406-1- Day 1: 1.5 hour postdose | 44.11 (78.5)
  ucb-100406-1- Day 1: 2 hours postdose | 52.59 (84.7)
  ucb-100406-1- Day 1: 3 hours postdose | 63.15 (83.9)
  ucb-100406-1- Day 1: 4 hours postdose | 73.57 (85.1)
  ucb-100406-1- Day 1: 6 hours postdose | 87.58 (85.6)
  ucb-100406-1- Day 1: 9 hours postdose | 91.89 (88.2)
  ucb-100406-1- Day 1: 12 hours postdose | 86.76 (88.6)
  ucb-100406-1- Day 1: 16 hours postdose | 78.88 (87.0)
  ucb-100406-1- Day 1: 24 hours postdose | 52.44 (86.2)
  ucb-100406-1- Day 1: 36 hours postdose | 22.54 (77.8)
  ucb-100406-1- Day 1: 48 hours postdose | 10.35 (72.1)
  ucb-100406-1- Day 1: 72 hours postdose | NA (NA) — Means, SDs and CVs were only calculated if at least 2/3 of the concentrations are above LLOQ.
  ucb107092-1- Day 1: Predose | NA (NA) — Means, SDs and CVs were only calculated if at least 2/3 of the concentrations are above LLOQ.
  ucb107092-1- Day 1: 0.25 hour postdose | NA (NA) — Means, SDs and CVs were only calculated if at least 2/3 of the concentrations are above LLOQ.
  ucb107092-1- Day 1: 0.5 hour postdose | NA (NA) — Means, SDs and CVs were only calculated if at least 2/3 of the concentrations are above LLOQ.
  ucb107092-1- Day 1: 1 hour postdose | 4.404 (62.9)
  ucb107092-1- Day 1: 1.5 hours postdose | 9.800 (32.1)
  ucb107092-1- Day 1: 2 hours postdose | 16.17 (22.6)
  ucb107092-1- Day 1: 3 hours postdose | 27.06 (18.3)
  ucb107092-1- Day 1: 4 hours postdose | 37.89 (22.1)
  ucb107092-1- Day 1: 6 hours postdose | 41.59 (16.3)
  ucb107092-1- Day 1: 9 hours postdose | 38.77 (25.1)
  ucb107092-1- Day 1: 12 hours postdose | 28.37 (20.8)
  ucb107092-1- Day 1: 16 hours postdose | 21.85 (22.0)
  ucb107092-1- Day 1: 24 hours postdose | 14.49 (28.7)
  ucb107092-1- Day 1: 36 hours postdose | 6.443 (23.4)
  ucb107092-1- Day 1: 48 hours postdose | 3.976 (29.0)
  ucb107092-1- Day 1: 72 hours postdose | NA (NA) — Means, SDs and CVs were only calculated if at least 2/3 of the concentrations are above LLOQ.

2. Primary Outcome: Plasma Concentration of BRV and Its Metabolites (Ucb-42145, Ucb-100406-1, ucb107092-1) After Multiple Dose
Time Frame: Predose on Day 5, 6, 7, 8, and 9; Day 10: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, and 72 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Brivaracetam: Participants received BRV 200 mg/day, orally from Day 5 to 9 and 100 mg on Day 10 in the multiple dose period.
Arm/Group | Brivaracetam
Number analyzed (Participants) | 12
ng/mL
  BRV- Day 5: Predose | NA (NA) — Means, SDs and CVs were only calculated if at least 2/3 of the concentrations are above LLOQ.
  BRV- Day 6: Predose | 1743 (33.6)
  BRV- Day 7: Predose | 1981 (36.3)
  BRV- Day 8: Predose | 1955 (38.4)
  BRV- Day 9: Predose | 1975 (41.7)
  BRV- Day 10: Predose | 1918 (34.2)
  BRV- Day 10: 0.25 hour postdose | 2888 (54.0)
  BRV- Day 10: 0.5 hour postdose | 4582 (45.6)
  BRV- Day 10: 1 hour postdose | 4448 (30.2)
  BRV- Day 10: 1.5 hour postdose | 4583 (21.5)
  BRV- Day 10: 2 hours postdose | 4421 (22.1)
  BRV- Day 10: 3 hours postdose | 4037 (23.3)
  BRV- Day 10: 4 hours postdose | 3671 (26.2)
  BRV- Day 10: 6 hours postdose | 2956 (26.7)
  BRV- Day 10: 9 hours postdose | 2241 (32.4)
  BRV- Day 10: 12 hours postdose | 1702 (38.4)
  BRV- Day 10: 16 hours postdose | 1185 (44.1)
  BRV- Day 10: 24 hours postdose | 614.7 (57.6)
  BRV- Day 10: 36 hours postdose | 216.1 (75.3)
  BRV- Day 10: 48 hours postdose | 93.68 (95.8)
  BRV- Day 10: 72 hours postdose | 17.75 (154)
  ucb-42145- Day 5: Predose | NA (NA) — Means, SDs and CVs were only calculated if at least 2/3 of the concentrations are above LLOQ.
  ucb-42145- Day 6: Predose | 153.6 (25.7)
  ucb-42145- Day 7: Predose | 185.8 (26.0)
  ucb-42145- Day 8: Predose | 181.1 (28.1)
  ucb-42145- Day 9: Predose | 193.1 (34.1)
  ucb-42145- Day 10: Predose | 166.6 (34.9)
  ucb-42145- Day 10: 0.25 hour postdose | 156.1 (38.3)
  ucb-42145- Day 10: 0.5 hour postdose | 177.0 (35.6)
  ucb-42145- Day 10: 1 hour postdose | 247.8 (34.5)
  ucb-42145- Day 10: 1.5 hour postdose | 265.2 (28.5)
  ucb-42145- Day 10: 2 hours postdose | 293.2 (26.2)
  ucb-42145- Day 10: 3 hours postdose | 357.2 (21.1)
  ucb-42145- Day 10: 4 hours postdose | 291.6 (27.0)
  ucb-42145- Day 10: 6 hours postdose | 199.9 (24.2)
  ucb-42145- Day 10: 9 hours postdose | 185.1 (28.4)
  ucb-42145- Day 10: 12 hours postdose | 123.7 (32.3)
  ucb-42145- Day 10: 16 hours postdose | 111.4 (33.7)
  ucb-42145- Day 10: 24 hours postdose | 54.35 (42.9)
  ucb-42145- Day 10: 36 hours postdose | 17.39 (59.5)
  ucb-42145- Day 10: 48 hours postdose | 9.114 (67.4)
  ucb-42145- Day 10: 72 hours postdose | NA (NA) — Means, SDs and CVs were only calculated if at least 2/3 of the concentrations are above LLOQ.
  ucb-100406-1- Day 5: Predose | NA (NA) — Means, SDs and CVs were only calculated if at least 2/3 of the concentrations are above LLOQ.
  ucb-100406-1- Day 6: Predose | 146.9 (78.9)
  ucb-100406-1- Day 7: Predose | 188.1 (75.4)
  ucb-100406-1- Day 8: Predose | 209.2 (72.1)
  ucb-100406-1- Day 9: Predose | 217.0 (71.3)
  ucb-100406-1- Day 10: Predose | 218.2 (71.8)
  ucb-100406-1- Day 10: 0.25 hour postdose | 221.2 (70.8)
  ucb-100406-1- Day 10: 0.5 hour postdose | 238.2 (67.6)
  ucb-100406-1- Day 10: 1 hour postdose | 243.9 (67.5)
  ucb-100406-1- Day 10: 1.5 hours postdose | 258.2 (70.9)
  ucb-100406-1- Day 10: 2 hours postdose | 249.9 (67.8)
  ucb-100406-1- Day 10: 3 hours postdose | 248.3 (69.1)
  ucb-100406-1- Day 10: 4 hours postdose | 254.3 (70.9)
  ucb-100406-1- Day 10: 6 hours postdose | 238.7 (68.7)
  ucb-100406-1- Day 10: 9 hours postdose | 229.0 (70.1)
  ucb-100406-1- Day 10: 12 hours postdose | 212.2 (76.0)
  ucb-100406-1- Day 10: 16 hours postdose | 171.7 (73.1)
  ucb-100406-1- Day 10: 24 hours postdose | 111.6 (72.8)
  ucb-100406-1- Day 10: 36 hours postdose | 41.71 (72.8)
  ucb-100406-1- Day 10: 48 hours postdose | 19.41 (66.7)
  ucb-100406-1- Day 10: 72 hours postdose | 2.771 (75.0)
  ucb107092-1- Day 5: Predose | NA (NA) — Means, SDs and CVs were only calculated if at least 2/3 of the concentrations are above LLOQ.
  ucb107092-1- Day 6: Predose | 51.71 (22.0)
  ucb107092-1- Day 7: Predose | 63.87 (27.2)
  ucb107092-1- Day 8: Predose | 65.14 (25.5)
  ucb107092-1- Day 9: Predose | 71.64 (23.3)
  ucb107092-1- Day 10: Predose | 68.47 (23.8)
  ucb107092-1- Day 10: 0.25 hour postdose | 62.74 (21.9)
  ucb107092-1- Day 10: 0.5 hour postdose | 63.76 (19.6)
  ucb107092-1- Day 10: 1 hour postdose | 65.20 (20.0)
  ucb107092-1- Day 10: 1.5 hours postdose | 68.84 (22.1)
  ucb107092-1- Day 10: 2 hours postdose | 71.72 (18.9)
  ucb107092-1- Day 10: 3 hours postdose | 82.18 (20.2)
  ucb107092-1- Day 10: 4 hours postdose | 84.04 (15.2)
  ucb107092-1- Day 10: 6 hours postdose | 80.87 (20.2)
  ucb107092-1- Day 10: 9 hours postdose | 69.25 (23.6)
  ucb107092-1- Day 10: 12 hours postdose | 52.96 (17.8)
  ucb107092-1- Day 10: 16 hours postdose | 42.69 (21.1)
  ucb107092-1- Day 10: 24 hours postdose | 28.57 (25.4)
  ucb107092-1- Day 10: 36 hours postdose | 13.15 (26.1)
  ucb107092-1- Day 10: 48 hours postdose | 8.580 (32.0)
  ucb107092-1- Day 10: 72 hours postdose | 3.380 (52.9)

3. Primary Outcome: Area Under the Plasma Concentration-time Curve From Zero to the Time of the Last Measured Concentration Above the Limit of Quantification (AUC(0-t)) of Brivaracetam for Single Dose
Description: AUC(0-t) was defined as the area under the plasma concentration-time curve from zero to the time of the last measured concentration above the limit of quantification.
Time Frame: Day 1: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, and 72 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanograms per milliliter (h*ng/mL)
Arm/Group | Brivaracetam
Number analyzed (Participants) | 12
hours*nanograms per milliliter (h*ng/mL) | 35730 (28.7)

4. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Brivaracetam for Single Dose
Description: Cmax was defined as the maximum observed plasma concentration.
Time Frame: Day 1: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, and 72 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Brivaracetam
Number analyzed (Participants) | 12
ng/mL | 3334 (22.2)

5. Primary Outcome: Area Under the Plasma Concentration-time Curve From 0 to 12 Hours at Steady State (AUC(0-12),ss) of Brivaracetam for Multiple Dose
Description: AUC(0-12),ss was defined as the area under the plasma concentration-time curve from 0 to 12 hours at steady state.
Time Frame: Day 10: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, and 12 hours postdose
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Brivaracetam
Number analyzed (Participants) | 12
h*ng/mL | 36760 (27.8)

6. Primary Outcome: Maximum Plasma Concentration at Steady State (Cmax,ss) of Brivaracetam for Multiple Dose
Description: Cmax,ss was defined as the maximum plasma concentration at steady state.
Time Frame: Day 10: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, and 72 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Brivaracetam
Number analyzed (Participants) | 12
ng/mL | 5215 (27.7)

7. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) During the Study
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. Treatment-emergent AEs (TEAEs) were defined as those events that start on or after the time of first investigational medicinal product (IMP) administration, or whose severity worsens on or after the date of first administration of the IMP.
Time Frame: From Baseline to the end of Safety Follow-up (approximately 6 weeks)
Population: The safety set consisted of all participants who received at least 1 dose of BRV.
Measure: Count of Participants; unit: Participants
Arm/Group | Brivaracetam
Number analyzed (Participants) | 12
Participants | 12

8. Secondary Outcome: Time to Reach Maximum Concentration (Tmax) of Brivaracetam, Ucb-42145, Ucb-100406-1 and ucb107092-1 in Plasma for Single Dose
Description: Tmax was defined as the time to reach maximum concentration. ucb-42145, ucb-100406-1, and ucb107092-1 are the metabolites of brivaracetam.
Time Frame: Day 1: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, and 72 hours postdose
Population: as for outcome 1
Measure: Median (Full Range); unit: hour
Arm/Group | Brivaracetam
Number analyzed (Participants) | 12
hour
  Brivaracetam | 1.000 [0.500 to 3.00]
  ucb-42145 | 3.000 [1.50 to 6.00]
  ucb-100406-1 | 9.000 [6.00 to 12.0]
  ucb107092-1 | 6.000 [4.00 to 9.00]

9. Secondary Outcome: Terminal Elimination Half-life (t1/2) of Brivaracetam, Ucb-42145, Ucb-100406-1 and ucb107092-1 in Plasma for Single Dose
Description: t1/2 was defined as the terminal elimination half-life. ucb-42145, ucb-100406-1, and ucb107092-1 are the metabolites of brivaracetam.
Time Frame: Day 1: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, and 72 hours postdose
Population: The PK-PPS consisted of all participants who were included in the safety set and also had a sufficient number of bioanalytical assessments to calculate reliable estimates for the primary PK parameters. Here, number analyzed signifies those who were evaluable at the prespecified categories only.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Brivaracetam
Number analyzed (Participants) | 12
hour
  Brivaracetam | 9.628 (2.229)
  ucb-42145 | 10.40 (2.716)
  ucb-100406-1 | 10.24 (1.696)
  ucb107092-1: number analyzed (Participants) | 10
  ucb107092-1 | 12.38 (1.019)

10. Secondary Outcome: Rate Constant of Elimination (λz) of Brivaracetam, Ucb-42145, Ucb-100406-1 and ucb107092-1 in Plasma for Single Dose
Description: λz was defined as the rate constant of elimination. ucb-42145, ucb-100406-1, and ucb107092-1 are the metabolites of brivaracetam.
Time Frame: Day 1: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, and 72 hours postdose
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour
Arm/Group | Brivaracetam
Number analyzed (Participants) | 12
1/hour
  Brivaracetam | 0.07370 (22.7)
  ucb-42145 | 0.06866 (25.3)
  ucb-100406-1 | 0.06847 (15.9)
  ucb107092-1: number analyzed (Participants) | 10
  ucb107092-1 | 0.05614 (8.10)

11. Secondary Outcome: Mean Residence Time (MRT) of Brivaracetam in Plasma for Single Dose
Description: MRT was defined as the mean residence time.
Time Frame: Day 1: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, and 72 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Brivaracetam
Number analyzed (Participants) | 12
hour | 13.02 (18.8)

12. Secondary Outcome: Area Under the Plasma Concentration-time Curve From 0 to Infinite Time (AUC) of Brivaracetam, Ucb-42145, Ucb-100406-1 and ucb107092-1 for Single Dose
Description: AUC was defined as the area under the plasma concentration-time curve from 0 to infinite time. ucb-42145, ucb-100406-1, and ucb107092-1 are the metabolites of brivaracetam.
Time Frame: Day 1: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, and 72 hours postdose
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Brivaracetam
Number analyzed (Participants) | 12
h*ng/mL
  Brivaracetam | 36000 (29.1)
  ucb-42145 | 2567 (25.4)
  ucb-100406-1 | 2530 (81.5)
  ucb107092-1: number analyzed (Participants) | 10
  ucb107092-1 | 878.2 (21.1)

13. Secondary Outcome: Apparent Total Body Clearance (CL/F) of Brivaracetam in Plasma for Single Dose
Description: CL/F was defined as the apparent total body clearance.
Time Frame: Day 1: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, and 72 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour (L/h)
Arm/Group | Brivaracetam
Number analyzed (Participants) | 12
Liter per hour (L/h) | 2.777 (29.1)

14. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of Brivaracetam in Plasma for Single Dose
Description: Vz/F was defined as the apparent volume of distribution.
Time Frame: Day 1: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, and 72 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Brivaracetam
Number analyzed (Participants) | 12
Liter | 37.69 (10.8)

15. Secondary Outcome: Cmax of Ucb-42145, Ucb-100406-1 and ucb107092-1 for Single Dose
Description: Cmax was defined as the maximum plasma concentration. ucb-42145, ucb-100406-1, and ucb107092-1 are the metabolites of brivaracetam.
Time Frame: Day 1: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, and 72 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Brivaracetam
Number analyzed (Participants) | 12
ng/mL
  ucb-42145 | 193.3 (27.7)
  ucb-100406-1 | 93.16 (88.0)
  ucb107092-1 | 43.18 (21.1)

16. Secondary Outcome: AUC (0-t) of Ucb-42145, Ucb-100406-1 and ucb107092-1 in Plasma for Single Dose
Description: AUC(0-t) was defined as the area under the plasma concentration-time curve from zero to the time of the last measured concentration above the limit of quantification. ucb-42145, ucb-100406-1, and ucb107092-1 are the metabolites of brivaracetam.
Time Frame: Day 1: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, and 72 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Brivaracetam
Number analyzed (Participants) | 12
h*ng/mL
  ucb-42145 | 2503 (25.4)
  ucb-100406-1 | 2423 (85.2)
  ucb107092-1 | 799.2 (21.1)

17. Secondary Outcome: Tmax of Brivaracetam, Ucb-42145, Ucb-100406-1 and ucb107092-1 in Plasma for Multiple Dose
Description: tmax is the time to reach maximum plasma concentration. ucb-42145, ucb-100406-1, and ucb107092-1 are the metabolites of brivaracetam.
Time Frame: Day 10: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, and 72 hours postdose
Population: as for outcome 1
Measure: Median (Full Range); unit: hour
Arm/Group | Brivaracetam
Number analyzed (Participants) | 12
hour
  Brivaracetam | 0.5000 [0.250 to 2.00]
  ucb-42145 | 3.000 [2.00 to 4.00]
  ucb-100406-1 | 1.500 [1.00 to 6.00]
  ucb107092-1 | 4.000 [0.00 to 6.02]

18. Secondary Outcome: t1/2 of Brivaracetam, Ucb-42145, Ucb-100406-1 and ucb107092-1 in Plasma for Multiple Dose
Description: t1/2 is the terminal elimination half-life. ucb-42145, ucb-100406-1, and ucb107092-1 are the metabolites of brivaracetam.
Time Frame: Day 10: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, and 72 hours postdose
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Brivaracetam
Number analyzed (Participants) | 12
hour
  Brivaracetam | 10.25 (1.749)
  ucb-42145 | 10.15 (2.198)
  ucb-100406-1 | 9.645 (1.067)
  ucb107092-1: number analyzed (Participants) | 7
  ucb107092-1 | 14.85 (2.334)

19. Secondary Outcome: λz of Brivaracetam, Ucb-42145, Ucb-100406-1 and ucb107092-1 in Plasma for Multiple Dose
Description: λz is the rate constant of elimination. ucb-42145, ucb-100406-1, and ucb107092-1 are the metabolites of brivaracetam.
Time Frame: Day 10: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, and 72 hours postdose
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour
Arm/Group | Brivaracetam
Number analyzed (Participants) | 12
1/hour
  Brivaracetam | 0.06860 (17.9)
  ucb-42145 | 0.06984 (22.4)
  ucb-100406-1 | 0.07228 (11.3)
  ucb107092-1: number analyzed (Participants) | 7
  ucb107092-1 | 0.04721 (16.5)

20. Secondary Outcome: Minimum Plasma Concentration at Steady State (Cmin,ss) of Brivaracetam in Plasma for Multiple Dose
Description: Cmin,ss is the minimum plasma concentration at steady state.
Time Frame: Day 10: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, and 72 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Brivaracetam
Number analyzed (Participants) | 12
ng/mL | 1696 (38.2)

21. Secondary Outcome: Average Plasma Concentration at Steady State (Cav,ss) of Brivaracetam in Plasma for Multiple Dose
Description: Cav,ss is the average plasma concentration at steady state.
Time Frame: Day 10: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, and 72 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Brivaracetam
Number analyzed (Participants) | 12
ng/mL | 3064 (27.8)

22. Secondary Outcome: Apparent Total Body Clearance at Steady State (CLss/F) of Brivaracetam in Plasma for Multiple Dose
Description: CLss/F is the apparent total body clearance at steady state.
Time Frame: Day 10: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, and 72 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Brivaracetam
Number analyzed (Participants) | 12
L/h | 2.720 (27.8)

23. Secondary Outcome: Vz/F of Brivaracetam in Plasma for Multiple Dose
Description: Vz/F is the apparent volume of distribution.
Time Frame: Day 10: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, and 72 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Brivaracetam
Number analyzed (Participants) | 12
Liter | 39.65 (14.8)

24. Secondary Outcome: Cmax,ss of Ucb-42145, Ucb-100406-1, and ucb107092-1 in Plasma for Multiple Dose
Description: Cmax,ss is the maximum plasma concentration at steady state. ucb-42145, ucb-100406-1, and ucb107092-1 are the metabolites of brivaracetam.
Time Frame: Day 10: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, and 72 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Brivaracetam
Number analyzed (Participants) | 12
ng/mL
  ucb-42145 | 357.9 (21.6)
  ucb-100406-1 | 264.8 (68.8)
  ucb107092-1 | 88.53 (16.1)

25. Secondary Outcome: Area Under the Curve From 0 to 12 Hours at Steady State (AUC(0-12),ss) of Ucb-42145, Ucb-100406-1 and ucb107092-1 in Plasma for Multiple Dose
Description: AUC(0-12),ss is the area under the curve from 0 to 12 hours at steady state. ucb-42145, ucb-100406-1, and ucb107092-1 are the metabolites of brivaracetam.
Time Frame: Day 10: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, and 12 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Brivaracetam
Number analyzed (Participants) | 12
h*ng/mL
  ucb-42145 | 2644 (23.5)
  ucb-100406-1 | 2844 (70.0)
  ucb107092-1 | 867.1 (18.3)

26. Secondary Outcome: Peak Trough Fluctuation (PTF) of Brivaracetam in Steady-state for Multiple Dose
Description: PTF was calculated as (Cmax,ss-Cmin,ss)/Cav,ss.
Time Frame: Day 10: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, and 72 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Brivaracetam
Number analyzed (Participants) | 12
ratio | 1.131 (24.2)

27. Secondary Outcome: Accumulation Ratio Calculated From AUC at Steady State and AUC After Single Dose (RAUC) of Brivaracetam for Multiple Dose
Description: Accumulation ratio (RAUC) was calculated as AUC(0-12),ss divided by AUC(0-12).
Time Frame: Day 10: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, and 12 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Brivaracetam
Number analyzed (Participants) | 12
ratio | 1.677 (12.6)

28. Secondary Outcome: Accumulation Ratio Calculated From Cmax at Steady State and Cmax After Single Dose (Rmax) of Brivaracetam for Multiple Dose
Description: Accumulation ratio (Rmax) was calculated as Cmax,ss divided by Cmax.
Time Frame: Day 10: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, and 72 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Brivaracetam
Number analyzed (Participants) | 12
ratio | 1.564 (30.4)

ADVERSE EVENTS:
Time Frame: From Day 1 to the end of Safety Follow-up (approximately 6 weeks)
Description: Treatment-emergent adverse events (TEAEs) are defined as adverse events (AEs) which have onset or worsening severity (relative to pre-treatment) after the first dose of BRV.
Arm/Group | Brivaracetam
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 12/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brivaracetam (N=12)
Neutrophilia (Blood and lymphatic system disorders) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 1 (2)
Ventricular extrasystoles (Cardiac disorders) | 1 (2)
Palpitations (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (5)
Asthenia (General disorders) | 3 (4)
Feeling drunk (General disorders) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 3 (4)
Blood pressure decreased (Investigations) | 1 (1)
Dizziness (Nervous system disorders) | 10 (15)
Somnolence (Nervous system disorders) | 7 (11)
Ataxia (Nervous system disorders) | 3 (3)
Haematuria (Renal and urinary disorders) | 1 (1)
Leukocyturia (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-01-08): https://cdn.clinicaltrials.gov/large-docs/40/NCT04882540/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-27): https://cdn.clinicaltrials.gov/large-docs/40/NCT04882540/SAP_001.pdf